CLINICAL TRIAL: NCT06330428
Title: Investigation of the Effect of Sexuality-Based Family Planning Education Given to Women Via Podcast on Contraceptive Method Selection and Sexual Life Quality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Zeynep Dilşah Karaçam Yılmaz, Lecturer, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MU-Ebe-ZDKY-02
Record Dates: First submitted 2024-03-12; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Contraception
Keywords: Family Planning; Contraceptive; Sexuality
MeSH Terms: conditions — Sexuality

STUDY DESIGN:
Intervention Model Description: One control group, one experimental group
Who Masked: Participant, Outcomes Assessor
Masking Description: The experimental group will receive sexuality-based family planning education via podcast and outcome assessment will be performed by an investigator who was blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Sexuality-based family planning education will be provided through podcasts.
  Interventions: Behavioral: Sexuality-Based Family Planning Education via Podcast
- Control group (No Intervention): Control

INTERVENTIONS:
Behavioral: Sexuality-Based Family Planning Education via Podcast — The training program is planned to consist of 5 modules. These trainings will be shared module by module on a daily basis through an application (Spotify) where podcasts are shared. These modules are as follows: 1. Sexual and Reproductive Health / Sexual Rights / Female-Male / Physiology of Sexual Functions, 2. Sexual Myths, 3. Contraceptive Methods-1, 4. Contraceptive Methods-2, 5. Sexually Transmitted Diseases / Safe Sexual Intercourse As a result of randomization, the links of the podcasts will be shared with the women in the experimental group one by one on a daily basis. Podcasts are planned to last an average of 10 minutes. This training content is planned for 5 days and the second tests will be applied by the researcher to the women who finish the podcasts. The 3rd tests will be applied 4 weeks after the second tests.
  Arms: Experimental group

SUMMARY:
In this study, it was aimed to examine the effect of Sexuality-Based Family Planning Education given to women of childbearing age via Podcast on contraceptive method selection and sexual life quality.

Accordingly, the hypotheses of the study are as follows:

Hypotheses of the Project H1: Sexuality-based family planning education via podcast has an effect on women's conscious and appropriate contraceptive method selection.

H2: Sexuality-based family planning education via podcast has a positive effect on women's sexual life quality.

H3: Sexuality-based family planning education via podcast has a positive effect on the quality of sexual life of women by increasing their level of contraceptive knowledge.

H4: Sexuality-based family planning education via podcast has a positive effect on women's attitudes towards family planning.

DETAILED DESCRIPTION:
The aim of this study was to examine the effect of sexuality-based family planning education given to women of childbearing age via podcast on contraceptive method selection and sexual life quality.

The study is planned to be conducted as a randomized controlled experimental study and women of childbearing age within the borders of Istanbul will be included in the study. The research will be conducted between November 2023 and May 2024 and a total of 176 women will be included in the study. The included women will be divided into two groups as experimental and control groups. Data will be collected by applying the Personal Information Form, Contraceptive Knowledge Rating Scale-Turkish Form (CKRA-TR), Sexual Quality of Life Scale-Woman (SQLS-W) and Family Planning Attitude Scale (FPAS). Women in the experimental group will be given sexuality-based family planning education consisting of 5 modules via podcasts. In addition, a brochure on family planning and education will be shared with the women in the experimental and control groups. The data obtained in the research will be entered into the database in IBM SPSS 29.0 (Statistical Package for the Social Sciences) program and all necessary statistical analyzes will be performed in the same program.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study,
* 15-49 years old,
* Does not have any physical or mental disability,
* At least primary school education,
* At least one sexual partner,
* Sexually active women will be included in the study.

Exclusion Criteria:

* Not sexually active in the last 4 weeks,
* Trained in the use of contraceptive methods,
* Being treated for any sexual dysfunction,
* Women with any psychiatric illness will be excluded from the study.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
Contraceptive Knowledge Assessment Scale-Turkish Form | Through study completion, an average of 6 months
  It will be used to measure contraception knowledge levels.

SECONDARY OUTCOMES:
Sexual Quality of Life Scale-Female | Through study completion, an average of 6 months
  It will be used to measure quality of life.

OTHER OUTCOMES:
Family Planning Attitudes Scale | Through study completion, an average of 6 months
  It will be used for the measurement of family planning attitudes.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zulu JM, Blystad A, Haaland MES, Michelo C, Haukanes H, Moland KM. Why teach sexuality education in school? Teacher discretion in implementing comprehensive sexuality education in rural Zambia. Int J Equity Health. 2019 Sep 27;18(1):116. doi: 10.1186/s12939-019-1023-1. PMID 31558168
- [Result] Calikoglu EO, Bilge Yerli E, Kavuncuoglu D, Yilmaz S, Kosan Z, Aras A. Use of Family Planning Methods and Influencing Factors Among Women in Erzurum. Med Sci Monit. 2018 Jul 19;24:5027-5034. doi: 10.12659/MSM.908388. PMID 30024863
- [Result] Slaymaker E, Scott RH, Palmer MJ, Palla L, Marston M, Gonsalves L, Say L, Wellings K. Trends in sexual activity and demand for and use of modern contraceptive methods in 74 countries: a retrospective analysis of nationally representative surveys. Lancet Glob Health. 2020 Apr;8(4):e567-e579. doi: 10.1016/S2214-109X(20)30060-7. Epub 2020 Mar 9. PMID 32164880